CLINICAL TRIAL: NCT03870035
Title: Role of Nesfatin-1 and Nicotinamide in Infertile Women With Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hassnaa Mahmoud Abd Elalem, Demonstrator, Assiut University
Other Study IDs: NESPCO
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-03

CONDITIONS: PCOS

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
evaluation of the potential role of circulating Nesfatin-1 and Nicotinamide in patients with polycystic ovary syndrome.

and detection the correlation between Nesfatin-1 and body mass index (BMI), Waist hip ratio (WHR), blood glucose, insulin, insulin resistance, lipid profiles, prolactin, LH, FSH, estrogen, progesterone, testosterone and dopamine.

DETAILED DESCRIPTION:
* Nesfatin-1 is an 82-amino acid polypeptide derived from the nucleobindin 2 (NUCB2) precursor proteins.
* It is a newly identified peptide. It is released from several tissues including forebrain, hindbrain, brainstem, spinal cord and adipose tissues.
* It plays an important role in hypothalamic pathways such as feeding inhibition, locomotion, stress modulation, thermogenesis, and reproduction.
* Several studies had demonstrated that nesfatin-1 associated with body mass index (BMI), insulin resistance and inflammatory response disorders.
* Polycystic ovary syndrome (PCOS) is one of the most common causes of infertility in women. It is characterized by hyperandrogenism, multiple ovarian cysts, oligomenorrhea/amenorrhea. Many mechanisms had been reported to be responsible for the pathophysiology of PCOS. The condition is thought to be interactions between hypothalamic-pituitary-ovarian, hypothalamic-pituitary-adrenal axis and metabolic disorders.
* The circulating level of nesfatin-1 in PCOS patients is controversial. Some studies reveal lower nesfatin-1 serum levels while others reveal higher level.
* Women with PCOS may have reduced dopamine production from the hypothalamus and elevated prolactin concentrations and this mechanism may be responsible for reproductive disorder.
* In PCOS, stimulation of reactive oxygen species (ROS) generation from mononuclear cells (MNCs) by hyperglycemia . The superoxide radical in particular is a ROS that is generated by the activity of membrane-bound nicotinamide adenine dinucleotide phosphate (NADPH) oxidase.
* Dopaminergic (DA) neurons are highly susceptible to ROS. DA is relatively unstable molecule and undergoes auto-oxidative metabolism in nigro striatal tract system, leading to ROS production. Nicotinamide can reduce hypothalamic dopamine in postnatal brains results in dopamine-deficient phenotypes. Nicotinamide prevents DA release induced by long-term perinatal asphyxia.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients in the age range 18 - 40 years old.
* Diagnosis of PCOS is based on the 2003 ESHRE/ASRM diagnostic criteria, according to which patients who had at least two of the following conditions are accepted as having PCOS:

  1. Oligo or anovulation, defined by the presence of oligomenorrhea or amenorrhea, confirmed by luteal progesterone and normal serum follicle stimulating hormone (FSH) levels (1.0-10.0 IU/L).
  2. Clinical hyperandrogenism signs which was defined as the presence of at least one of the following three features: hirsutism, acne, and androgenic alopecia. Biochemical hyperandrogenism was defined as a serum testosterone (T) level >60 ng/dL (>2.08 nmol/L).
  3. PCOS manifestation was defined as the presence of >12 unilateral follicles 2-9 mm in size on the ovary or having the least unilateral ovary volume of 10 cm3 by ultrasonography (the measurement was performed when there was no follicle >10 mm). Ovarian volume was calculated by the formula [0.5× ovarian length × thickness × width]. In the case of transabdominal ultrasonography, the presence of at least 10 unilateral antral follicles was required.

Exclusion Criteria:

* Patients (age <18 or > 40years),
* Other endocrinology diseases as diabetes mellitus or thyroid disorders, Brain disorders as pituitary adenoma or tumour or brain tumours or masses,
* Chronic diseases such as cardiovascular, hepatic, hematologic, chronic renal failure, hypertension, and cancer,
* Use of oral contraceptives, antiandrogenics, glucocorticoids, antihypertensives, antidiabetics and anti-obesity drugs as well as the cigarettes, alcohol, and patients unwilling to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: The PCOS patients included in this study will be selected from out patient's clinic of the department of Obstetrics and Gynaecology at Assiut university hospital, Assiut, Egypt, during one year after the study begins. Informed consent will be obtained from each patient before the examination after explaining the aim of the study to each participant, and the study will be approved by the ethical committee of our institution. The gathered demographic information and complete data will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate role of nesfatin-1, nicotinamide and dopamine plasma levels in patients with polycystic ovary syndrome. | Baseline
  Measurement of the circulating plasma levels of nesfatin-1, nicotinamide, and dopamine using the corresponding enzyme linked immunosorbent assay (ELISA) kit

SECONDARY OUTCOMES:
Detect the correlation between nesfatin-1, nicotinamide and dopamine plasma levels and BMI, WHR, insulin resistance, lipid profile, prolactin, LH, FSH, testosterone, estradiol, progesterone. | Baseline
  Determination of homeostasis model of insulin resistance (HOMA-IR): Serum insulin concentration measured using a human insulin ELISA kit. The insulin resistance assessed by homeostasis model assessment estimate of insulin resistance (HOMA-IR):
  HOMA-IR = Fasting insulin (IU/ml) × Fasting glucose (mmol/L)/22.5
  Determination of lipid profile: Total cholesterol, triglycerides and high density lipoprotein-cholesterol measured by the corresponding kit. Whereas, low density lipoprotein-cholesterol concentrations estimated according to the formula: LDL-cholesterol = Total cholesterol - [HDL-cholesterol + TG/5)].
  routine investigation as hormonal assay as estradiol, progesterone, testosterone, prolactin, FSH, LH
  Measurement of weight, height, hip circumference, waist circumference

CONTACTS AND LOCATIONS:
Overall Officials: Hayam G Sayyed, Professor, Study Director — Assiut University

REFERENCES:
- [Result] Slivka A, Cohen G. Hydroxyl radical attack on dopamine. J Biol Chem. 1985 Dec 15;260(29):15466-72. PMID 2999117
- [Result] Oh-I S, Shimizu H, Satoh T, Okada S, Adachi S, Inoue K, Eguchi H, Yamamoto M, Imaki T, Hashimoto K, Tsuchiya T, Monden T, Horiguchi K, Yamada M, Mori M. Identification of nesfatin-1 as a satiety molecule in the hypothalamus. Nature. 2006 Oct 12;443(7112):709-12. doi: 10.1038/nature05162. Epub 2006 Oct 1. PMID 17036007
- [Result] Sahin FK, Sahin SB, Ural UM, Cure MC, Senturk S, Tekin YB, Balik G, Cure E, Yuce S, Kirbas A. Nesfatin-1 and Vitamin D levels may be associated with systolic and diastolic blood pressure values and hearth rate in polycystic ovary syndrome. Bosn J Basic Med Sci. 2015 Jul 9;15(3):57-63. doi: 10.17305/bjbms.2015.432. PMID 26295295
- [Result] Yosten GL, Samson WK. The anorexigenic and hypertensive effects of nesfatin-1 are reversed by pretreatment with an oxytocin receptor antagonist. Am J Physiol Regul Integr Comp Physiol. 2010 Jun;298(6):R1642-7. doi: 10.1152/ajpregu.00804.2009. Epub 2010 Mar 24. PMID 20335376
- [Result] Kostal M, Tosner J. The influence of latent hyperprolactinaemia on the levels of LH, FSH, E2 and T in the midfollicular phase of the cycle. Arch Gynecol Obstet. 1997;259(2):65-8. PMID 9059746